CLINICAL TRIAL: NCT04778449
Title: Quality of Life, Lifestyle, and Psychosocial Factors in Patients With Melanoma
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0336; NCI-2020-08200 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA15-0336 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-19; First posted 2021-03-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cutaneous Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire, medical chart review): Patients complete a maximum of 3 paper or electronic questionnaires over 30 minutes within 2 weeks of presentation to MD Anderson, new diagnosis of melanoma, and/or initiating a new treatment, within 2 weeks of first restaging, and within 2 weeks of the end of treatment. Patients may complete an additional paper or electronic dietary questionnaire over 10 minutes for 3 days (30 minutes total) or a phone-based dietary recall. Patients who start a new treatment of interest may repeat the questionnaires at the same time points. Patients' medical records are also reviewed.
  Interventions: Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Medical Chart Review — Medical charts are reviewed
  Other Names: Chart Review
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the extent to which lifestyle factors including mental health, social support, diet, and exercise are associated with quality of life and melanoma patient outcomes. Knowledge gained from this study may be used to guide the design of prospective clinical trials of lifestyle interventions to improve the outcomes of melanoma patients and assist doctors in counseling their patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collect systematic data on mental health, quality of life (QOL), social support, diet, and exercise behaviors in melanoma patients.

II. Examine whether psychosocial factors and lifestyle are associated with clinical outcomes in melanoma patients.

III. Examine the association between lifestyle and psychosocial factors and tissue and blood biomarkers in melanoma patients.

IV. Examine whether psychosocial factors and lifestyle are associated with QOL adjustment in melanoma patients.

OUTLINE:

Patients complete a maximum of 3 paper or electronic questionnaires over 30 minutes within 2 weeks of presentation to MD Anderson, new diagnosis of melanoma, and/or initiating a new treatment, within 2 weeks of first restaging, and within 2 weeks of the end of treatment. Patients may complete an additional paper or electronic dietary questionnaire over 10 minutes for 3 days (30 minutes total) or a phone-based dietary recall. Patients who start a new treatment of interest may repeat the questionnaires at the same time points. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma, precursor lesions, and associated cutaneous pathology
* Able to read and understand English
* Willing to complete an online or paper survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma, precursor lesions, and associated cutaneous pathology
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-08-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression/distress | Up to 10 years
  Will be assessed using the Centers for Epidemiologic Studies - Depression. Lifetime history of Major Depressive Disorder (MDD) will be measured using the two cardinal items from the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-IV Disorder. Multivariate methods, including repeated measures analyses, will be employed to further explore the potential changes in the measures over time.
Change in anxiety | Up to 10 years
  Will be assessed using the Speilberger State/Trait Anxiety Inventory. Multivariate methods, including repeated measures analyses, will be employed to further explore the potential changes in the measures over time.
Change in cancer-related symptoms | Up to 10 years
  Will be assessed using the MD Anderson Symptom Inventory. Multivariate methods, including repeated measures analyses, will be employed to further explore the potential changes in the measures over time.
Change in social support | Up to 10 years
  Will be assessed using the 24-item Social Provisions Scale. Multivariate methods, including repeated measures analyses, will be employed to further explore the potential changes in the measures over time.
Change in general eating habits | Up to 10 years
  Will be assessed using the National Cancer Institute National Health and Nutrition Examination Survey Dietary Screener Questionnaire, and optionally, the National Institutes of Health Automated Self-Administered 24-hour.
Change in physical activity | Up to 10 years
  Will be assessed using the Godin Leisure -Time Exercise Questionnaire. Multivariate methods, including repeated measures analyses, will be employed to further explore the potential changes in the measures over time.
Associations between mental health, social support, diet and exercise behaviors, and quality of life and demographic variables | Up to 10 years
  Will be evaluated using Pearson's product moment correlation coefficients together with scatterplots where appropriate.
Effect of diet, physical activity, depressive symptoms, distress, lifetime MDD, and social support on progression free survival | Up to 10 years
  Will be evaluated using Pearson's product moment correlation coefficients together with scatterplots where appropriate.
Effect of diet, physical activity, depressive symptoms, distress, lifetime MDD, and social support on cancer mortality | Up to 10 years
  Will be evaluated using Pearson's product moment correlation coefficients together with scatterplots where appropriate.
Response to treatment | Up to 10 years
  Logistic regression models will be used to measure the association of diet, physical activity, diet, depressive symptoms, distress, lifetime MDD, and social support and response to treatment at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L McQuade, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org